CLINICAL TRIAL: NCT00443443
Title: A Long-Term Study of the Safety of Rituxan in Patients With Rheumatoid Arthritis After an Inadequate Response to Previous Anti-TNF Therapy (SUNSTONE)
Brief Title: A Study of the Safety of Rituxan in Patients With Rheumatoid Arthritis After an Inadequate Response to Previous Anti-TNF Therapy (SUNSTONE)
Acronym: SUNSTONE
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: U3839g; BIIB
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rituximab; RA; Sunstone; anti-TNF; Rituxan
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This is an observational study designed to follow patients with RA who have had an inadequate response to one or more anti-TNF therapies and who will receive Rituxan. Approximately 1000 patients in the United States with RA who have had an inadequate response to anti-TNF therapies and who will receive Rituxan therapy will be recruited. There is no protocol mandated treatment assignment in this study. Patients will be evaluated and treated according to their physician's standard practice and discretion.

ELIGIBILITY:
Inclusion Criteria:

* No prior use of Rituxan (except if received within 8 weeks of screening)
* Signed Informed Consent Form
* Age ≥ 18 years
* Diagnosis of RA
* Inadequate response to one or more anti-TNF therapies

Exclusion Criteria:

* Have known hypersensitivity to any component of a humanized or murine monoclonal antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RA who have had an inadequate response to one or more anti-TNF therapies
Sampling Method: Non-Probability Sample
Enrollment: 1026 (Actual)
Dates: Start 2007-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Swati Tole, M.D., M.S., Study Director — Genentech, Inc.
Locations (193):
- United States (192):
  - Rheumatology Associates, PC, Birmingham, Alabama
  - Rheumatology Associates of N. AL, P.C., Huntsville, Alabama
  - Clinic for Rheumatic Diseases - Research Department, Tuscaloosa, Alabama
  - Arizona Arthritis and Rheumatology Research, PLLC, Paradise Valley, Arizona
  - Phoenix Rheumatology Specialists, Ltd., Phoenix, Arizona
  - Advanced Arthritis Care & Research, Scottsdale, Arizona
  - The Arthritis Center of the Ozarks, Fayetteville, Arkansas
  - Investigational Site, Covina, California
  - Arthritis Medical Clinic of North County, Inc., Escondido, California
  - Solano Regional Medical Group, Fairfield, California
  - Clinical Trials of St. Jude Heritage Medical Group, Fullerton, California
  - Investigational Site, Hemet, California
  - Allergy and Rheumatology Medical Clinic, Inc, La Jolla, California
  - Investigational Site, La Mesa, California
  - Arthritis Center of Southern Orange County, Laguna Hills, California
  - VA Loma Linda Healthcare System, Loma Linda, California
  - Valerius Medical Group and Research Center of Greater Long Beach, Inc., Long Beach, California
  - Beverly Medical Associates, Los Angeles, California
  - Investigational Site, Los Angeles, California
  - Samaritan Center for Medical Research, Medical Group, Los Gatos, California
  - Mission Internal Medical Group- Rheumatology Division, Mission Viejo, California
  - Investigational Site, Newport Beach, California
  - Rheumatology Associates, North Hollywood, California
  - Desert Medical Advances, Palm Desert, California
  - Arthritis Medical Clinic, Riverside, California
  - East Bay Rheumatology Medical Group, San Leandro, California
  - Pacific Arthritis Center Medical Group, Santa Maria, California
  - Healthcare Partners Medical Group, Torrance, California
  - Investigational Site, Torrance, California
  - Desert Valley Medical Group, Victorville, California
  - Investigational Site, Visalia, California
  - Agilence Arthritis & Osteoporosis Medical Center, Inc., Whittier, California
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Medical and Research Center, Denver, Colorado
  - Arthritis and Rheumatology Clinic of Northern Colorado, LLC, Fort Collins, Colorado
  - Greeley Medical Clinic, Greeley, Colorado
  - Colorado Center for Arthritis and Osteoporosis, Longmont, Colorado
  - Investigational Site, Bridgeport, Connecticut
  - Clinical Research Center of CT/NY, Danbury, Connecticut
  - University of CT Health Center, Farmington, Connecticut
  - The William W. Backus Hospital, Norwich, Connecticut
  - Delaware Arthritis & Osteoporosis Center, Newark, Delaware
  - VAMC, Washington D.C., District of Columbia
  - RASF- Clinical Research, Boca Raton, Florida
  - Countryside Arthritis Center, Clearwater, Florida
  - MIMA Century Research Associates, Melbourne, Florida
  - Investigational Site, Naples, Florida
  - Naples Medical Center, Naples, Florida
  - Arthritis & Osteoporosis Treatment Research Center, Inc., North Miami Beach, Florida
  - Arthritis & Osteoporosis Treatment Center, P.A., Orange Park, Florida
  - Investigational Site, Orlando, Florida
  - Rheumatology Associates of Central Florida, PA, Orlando, Florida
  - Suncoast Medical Clinic, LLC, St. Petersburg, Florida
  - Brookshire Rheumatology & Wellness Center, Tampa, Florida
  - Lake Rheumatology, Tavares, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Georgia Internal Medicine Associates, PA, Austell, Georgia
  - Arthritis Center of North Georgia, Gainesville, Georgia
  - North Georgia Rheumatology Group, PC, Lawrenceville, Georgia
  - Middle Georgia Arthritis Center, Macon, Georgia
  - Arthritis and Osteoporosis Center of South Georgia, Tifton, Georgia
  - Valdosta Specialty Clinic, Valdosta, Georgia
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Northern Illinois Research Associates, DeKalb, Illinois
  - Prairie Rheumatology Associates, S.C., Joliet, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Arthritis Care Center, PC, Moline, Illinois
  - Rockford Orthopedic Associates, Rockford, Illinois
  - Integrative Pain Medicine, Schaumburg, Illinois
  - Physicians Clinic Of Iowa, Cedar Rapids, Iowa
  - Mercy Arthritis and Osteoporosis Center, Des Moines, Iowa
  - Medical Associates Clinic PC, Dubuque, Iowa
  - Arthritis and Rheumatology Clinics of Kansas, Wichita, Kansas
  - Ashland Arthritis Center, Ashland, Kentucky
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Rheumatology Associates, Louisville, Kentucky
  - Lafayette Arthritis & Endocrine Clinic, Lafayette, Louisiana
  - Investigational Site, Lewiston, Maine
  - Investigational Site, Baltimore, Maryland
  - Rheumatology Associates of Baltimore, Baltimore, Maryland
  - Maryland Arthritis Care Specialists, Ellicott City, Maryland
  - Northampton Internal Medicine Associates, P.C., Florence, Massachusetts
  - Ann Arbor Rheumatology, Ann Arbor, Michigan
  - Associated Internal Medicine Specialists, P.C., Battle Creek, Michigan
  - Michigan Arthritis Research Center, Brighton, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Investigational Site, East Lansing, Michigan
  - Lansing Rheumatology, PLLC, East Lansing, Michigan
  - Arthritis Education and Treatment Center, PLLC, Grand Rapids, Michigan
  - Cascades Rheumatology, Jackson, Michigan
  - Shores Rheumatology P.C., Saint Clair Shores, Michigan
  - Southwest MI Rheumatology Center, Saint Joseph, Michigan
  - Whiteside Institute for Clinical Research, Duluth, Minnesota
  - St. Paul Rheumatology PA, Eagan, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Arthritis and Osteoporosis Treatment and Research Center, Flowood, Mississippi
  - Arthritis Associates, PLLC, Hattiesburg, Mississippi
  - Investigational Site, Pascagoula, Mississippi
  - NMMC-IMA Tupelo, Tupelo, Mississippi
  - Cape Girardeau Physician Associates, Cape Girardeau, Missouri
  - North County Medicine & Rheumatology, Florissant, Missouri
  - Hannibal Clinic, Hannibal, Missouri
  - Rheumatology and Internal Medicine Associates of West County, P.C., St Louis, Missouri
  - The Arthritis & Osteoporosis Center, P.C., Billings, Montana
  - Osteoporosis and Arthritis Center, Henderson, Nevada
  - Investigational Site, Las Vegas, Nevada
  - Allergy and Arthritis Associates, Dover, New Jersey
  - Arthritis and Osteoporosis Associates, PA, Manalapan, New Jersey
  - Rheumatology and Arthritis Associates, P.C., Medford, New Jersey
  - Investigational Site, Midland Park, New Jersey
  - Investigational Site, Ridgewood, New Jersey
  - Albuquerque Rehabilitation and Rheumatology, PC, Albuquerque, New Mexico
  - Arthritis and Osteoporosis Associates, Las Cruces, New Mexico
  - Investigational Site, Los Alamos, New Mexico
  - The Center for Rheumatology, LLP, Albany, New York
  - Investigational Site, Garden City, New York
  - Bay Rheumatology PC, Great Neck, New York
  - Rheumatology Consultants, LLP, Hewlett, New York
  - Hospital for Special Surgery, New York, New York
  - Research Across America - New York, New York, New York
  - Allergy, Immunology, Rheumatology Clinical Group, Rochester, New York
  - Arthritis Center of Rochester, Rochester, New York
  - Rheumatology Associates of Long Island, Smithtown, New York
  - Arthritis Health Associates, Syracuse, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - UNC Thurston Arthritis Research Center, Chapel Hill, North Carolina
  - Joint and Muscle Medical Care, Charlotte, North Carolina
  - Arthritis Clinic & Carolina Bone & Joint, Charlotte, North Carolina
  - LaFayette Clinic, PA, Fayetteville, North Carolina
  - Physicians East, Greenville, North Carolina
  - Carolina Arthritis Associates, P.A., Wilmington, North Carolina
  - Medcenter One, Bismarck, North Dakota
  - Children's Hospital Medical Center of Akron d/b/a Akron Children's Hospital, Akron, Ohio
  - Crystal Arthritis Center Inc., Akron, Ohio
  - Arthritis Clinic of Stark County, Inc., Canton, Ohio
  - Arthritis Center, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Columbus Arthritis Center, Columbus, Ohio
  - Dayton Outpatient Center, Dayton, Ohio
  - Southwest Rheumatology and Research Goup, LLC, Middleburg Heights, Ohio
  - University Hospitals Case Medical Center, Orange, Ohio
  - Arthritis Associates of Northwest Ohio, Inc., Toledo, Ohio
  - Physicians Building Group, LLP, Salem, Oregon
  - Rheumatology Associates, LTD, Colmar, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Lebanon Internal Medicine Associates, P.C., Lebanon, Pennsylvania
  - Arthritis & Rheumatic Disease Associates, LLC, Monroeville, Pennsylvania
  - Einstein Arthritis Center, Philadelphia, Pennsylvania
  - The Arthritis Group, Philadelphia, Pennsylvania
  - Investigational Site, West Chester, Pennsylvania
  - Clinical Research Center of Reading, LLP, West Reading, Pennsylvania
  - Allegheny North Arthritis Center, PC, Wexford, Pennsylvania
  - Investigational Site, Wynnewood, Pennsylvania
  - Rheumatology Associates, Charleston, South Carolina
  - Carolina Healthcare, Florence, South Carolina
  - Carolina Rheumatology and Neurology Associates, PC, Myrtle Beach, South Carolina
  - Strand Physician Specialists PA DBA Carolina Health Specialists, Myrtle Beach, South Carolina
  - Acme Research, L.L.C., Orangeburg, South Carolina
  - Carolina Medical Affiliates, Spartanburg, South Carolina
  - CMC Speciality Group, Crossville, Tennessee
  - Rheumatology Consultants PLLC, Knoxville, Tennessee
  - Heritage Medical Associates, P.C., Nashville, Tennessee
  - Abilene Arthritis Center, Abilene, Texas
  - Investigational Site, Bedford, Texas
  - Arthritis Clinic, Carrollton, Texas
  - Investigational Site, Dallas, Texas
  - Presbyterian Hospital Dallas Arthritis Consultation Center, Dallas, Texas
  - Rheumatology Associates, Dallas, Texas
  - Rheumatic Disease Clinic of Houston, Houston, Texas
  - Evergreen Clinical Research, LLC, Houston, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Arthritis & Osteoporosis Center, Midland, Texas
  - Center for Arthritis and Rheumatic Diseases, San Antonio, Texas
  - Arthritis and Rheumatic Disease Associates, PC, Burke, Virginia
  - Center for Arthritis & Rheumatic Diseases, P.C., Chesapeake, Virginia
  - NDC Medical Center, Norfolk, Virginia
  - Investigational Site, Portsmouth, Virginia
  - Northern Virginia Center for Arthritis, Reston, Virginia
  - Premier HealthCare Associates Inc., Richmond, Virginia
  - Arthritis and Rheumatic Diseases, PC, Williamsburg, Virginia
  - Investigational Site, Kirkland, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Investigational Site, Tacoma, Washington
  - Rheumatology & Pulmonary Clinic, Beckley, West Virginia
  - Rural Outreach Arthritis Center, Martinsburg, West Virginia
  - Rheumatic Disease Center, Glendale, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Gundersen Clinic, Ltd., Onalaska, Wisconsin
- San Juan Arthritis and Research Center, Inc., San Juan, Puerto Rico